CLINICAL TRIAL: NCT04121468
Title: A Phase I Double Blind Study of Metformin Acting on Endogenous Neural Progenitor Cells in Children and Young Adults With Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Queen's University (Other); Ontario Institute for Regenerative Medicine (Unknown); Unity Health Toronto (Other); Stem Cell Network (Other); Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Senior Associate Scientist, Division of Neuroscience and Mental Health, SickKids Research Institute, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000059119
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis (MS)
Keywords: remyelination; youth; white matter; neural precursor cells; clinical trial; metformin
MeSH Terms: conditions — Multiple Sclerosis | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Multiple baseline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Other): Placebo for 3 months at dose of 500 mg/m2/day po (to be rounded) given in 1 or 2 divided doses for one week and if there are no side effects increased to 1000 mg/m2/day po given in 2 divided doses up to a maximum dose of 2000 mg/day.
  Metformin for 9 months at dose of 500 mg/m2/day po (to be rounded) given in 1 or 2 divided doses for one week and if there are no side effects increased to 1000 mg/m2/day po given in 2 divided doses up to a maximum dose of 2000 mg/day.
  Interventions: Drug: Metformin; Other: Placebo
- Group B (Other): Placebo for 6 months at dose of 500 mg/m2/day po (to be rounded) given in 1 or 2 divided doses for one week and if there are no side effects increased to 1000 mg/m2/day po given in 2 divided doses up to a maximum dose of 2000 mg/day.
  Metformin for 6 months at dose of 500 mg/m2/day po (to be rounded) given in 1 or 2 divided doses for one week and if there are no side effects increased to 1000 mg/m2/day po given in 2 divided doses up to a maximum dose of 2000 mg/day.
  Interventions: Drug: Metformin; Other: Placebo
- Group C (Other): Placebo for 9 months at dose of 500 mg/m2/day po (to be rounded) given in 1 or 2 divided doses for one week and if there are no side effects increased to 1000 mg/m2/day po given in 2 divided doses up to a maximum dose of 2000 mg/day.
  Metformin for 3 months at dose of 500 mg/m2/day po (to be rounded) given in 1 or 2 divided doses for one week and if there are no side effects increased to 1000 mg/m2/day po given in 2 divided doses up to a maximum dose of 2000 mg/day.
  Interventions: Drug: Metformin; Other: Placebo

INTERVENTIONS:
Drug: Metformin — Each tablet contains 500mg of metformin hydrochloride
  Other Names: Glucophage
Other: Placebo — Each tablet contains no active drug ingredient

SUMMARY:
A randomized multiple baseline feasibility trial where participants will start taking metformin at one of 3 randomly determined points (3-months, 6-months or 9 months) during the 12-month trial. All subjects will be on a daily dose of metformin for a minimum of 3 months and a maximum of 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of MS with anterior visual pathway involvement and longer than 6 months after presentation with ON or an acute demyelinating event/relapse
* Age 10 year to 25 years and 11 months
* Latency delay > 115 milliseconds on baseline full-field transient pattern reversal VEP in at least one eye (electrophysiological evidence of demyelination) or > 10 milliseconds difference between eyes, or Retinal Nerve Fiber Layer (RNFL) thickness on OCT of < 90 µm in at least one eye or an inter-eye difference in the RNFL of 10 µm or more
* Retinal Nerve Fiber Layer (RNFL) Thickness on baseline OCT ≥60 µm
* If on an MS disease-modifying therapy, no changes in the therapeutic agent or dosing in the 6 months prior to study initiation
* No significant renal or liver abnormalities
* Expanded Disability Status Scale (EDSS) 0-6.0 (inclusive)
* Has either English as his or her native language or English comprehension needed to complete the neuropsychological testing
* Meet criteria for adequate organ function requirements as described below:

Adequate renal function defined as:

Creatinine clearance or radioisotope glomerular filtration rate (GFR) > 70 mL/min/1.73 m2 or serum creatinine based on age/gender as follows:

Range Serum Creatinine Level (µmol/L): Age 5 to <12 years (male)=25-50, Age 5 to <12 years (female)=25-50; Age 12 to <15 years (male)=37-67, Age 12 to <15 years (female)=37-67; Age 15 to <19 years (male)=51-89, Age 15 to <19 years (female)=40-69; Age ≥19 years (male)=58-110; Age ≥19 years (female)=46-92

Adequate liver function defined as:

Total bilirubin < 1.5 x upper limit of normal (ULN) for age SGOT (AST) or SGPT (ALT) < 1.5 x upper limit of normal (ULN) for age

Exclusion Criteria:

* A history of retinal pathology (major ophthalmologic disease / concomitant ophthalmologic disorders)
* Unstable and/or insulin-dependent (Type 1) diabetes, metabolic acidosis and/or lactic acidosis
* History of unexplained hypoglycemia (<2.8 mmol/L)
* Already on metformin
* Concomitant use of any other putative remyelinating therapy as determined by the Principal/Qualified Investigator
* Treatment for an acute attack with corticosteroids within 30 days prior to screening / relapse within 30 days prior to screening
* Concomitant use of insulin
* Concomitant use of any drugs that are listed to have drug-drug interactions with metformin (i.e. calcium channel blockers, diuretics, etc.) as determined by Principal/Qualified Investigator
* Lactate levels > 1.5x upper limit of normal
* Pregnancy

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (safety and tolerability) | 3 years
Number of patients who were approached to participate, declined participation and consented to participate (recruitment) | 3 years
Proportion of patients who completed each visit within the trial (retention) | 3 years
Proportion of patients who completed each of the outcome measures at the appropriate time points (adherence with outcome measures) | 3 years
Number of patients enrolled in the study compared to the number of patients who were able to complete study measures (tolerability with outcome measures) | 3 years

SECONDARY OUTCOMES:
Optical Coherence Tomography (OCT) - Retinal Nerve Fiber Layer Thickness | 3 years
Optical Coherence Tomography (OCT) - Ganglion Cell Inner Plexiform Layer Thickness | 3 years
Optical Coherence Tomography (OCT) - Optic Nerve Head Volume | 3 years
Visual Evoked Potentials (VEP) - p100 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: E. Ann Yeh, MA, MD, FRCPC, Dip ABPN, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No